CLINICAL TRIAL: NCT01884688
Title: A Phase II Study of Autologous Expanded Natural Killer Cell Therapy for Asymptomatic Multiple Myeloma
Brief Title: UARK 2013-05 A Study of Autologous Expanded Natural Killer Cell Therapy for Asymptomatic Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 138826
Record Dates: First submitted 2013-06-10; First posted 2013-06-24 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Asymptomatic Multiple Myeloma
Keywords: Asymptomatic Multiple Myeloma; Auto-ENK Cell Therapy; Natural Killer Cells
MeSH Terms: conditions — Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ENK Cell Infusion (Experimental): Expanded Natural Killer Cell Infusion
  Interventions: Drug: ENK Cell Infusion

INTERVENTIONS:
Drug: ENK Cell Infusion — Day 0(1 dose) ENK Cell Infusion Day 0 to + 12 (13 doses) Aldesleukin (IL2), 3x10 IU
  Other Names: Auto-ENK Cell Therapy

SUMMARY:
The purpose of this study is to determine the safety and in vivo persistence and expansion of autologous and expansion of autologous, ex vivo expanded-natural killer(ENK) cells.

DETAILED DESCRIPTION:
To determine whether significant in vivo expansion of auto-ENK cells occurs, defined as a > 4 fold increase in absolute cluster of differentiation 3(CD3)-cluster of differentiation 56 (CD56+) NK cell count/blood 7 days after infusion over the pre-study baseline level and the safety of the ENK cell therapy in research participants with high-risk asymptomatic multiple myeloma (AMM) defined as gene expression profile (GEP) 70 gene score>-0.26.

ELIGIBILITY:
Inclusion Criteria:

* The study population will be participants with AMM being seen at Myeloma Institute for Research and Therapy (MIRT), and under continuing followup with standard clinical care testing .
* Participants must have a diagnosis of AMM as defined in Staging Criteria (Section 3.0) and GEP-70 score >-0.26.
* Participant (male or female) from any race or ethnicity must be at least 18 years of age and not older than 75 years of age at the time of registration.
* Participants must have a performance status of 0 - 2 by Zubrod criteria
* Participants must have signed an Institutional Review Board (IRB)-approved informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization form.
* Must be fit to undergo leukapheresis for ENK cell generation as determined by PI.
* Must be a suitable candidate for insertion of apheresis catheter. Participants with unusual anatomy or vascular anomalies preventing insertion of apheresis catheter will not qualify.
* Patients must have previous test results indicating adequate pulmonary function studies (PFT) > 50% of predicted on mechanical aspects (FEV1, forced vital capacity(FVC), etc) and diffusion capacity (DLCO) > 50% of predicted.

Exclusion Criteria:

* Participants must not have received prior treatment for their disease. Prior use of bisphosphonates is permitted.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 2 years.
* May not have history of poorly-controlled hypertension, diabetes mellitus, or any other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol or could be considered to be an exclusion criterion deemed by the PI.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy test documented within 10 to 14 days of enrollment. Women/men of reproductive potential may not participate unless they have either agreed to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg,calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.) OR begin TWO reliable methods of birth control: 1 highly effective method and 1 additional effective method AT THE SAME TIME, at least 28 days before starting study treatment through 30 days after the last dose of study treatment.
* Serologic evaluation will be used to assess exposure to syphilis, West Nile Virus, Chagas, cytomegalovirus (CMV), Immunoglobulin G (IgG), hepatitis B, and C, HIV I and II, and human t cell lymphoma virus (HTLV) I/II. Participants may not be hepatitis B or C (+) unless positive due to previous vaccination or positive but has received therapy and is negative for hepatitis B or C by rapid test polymerase chain reaction (RT-PCR). An HIV-I/II(+) and HTLV-1/II (+) participant will be rejected on medical grounds. Participants serologically positive for syphilis, West Nile Virus, Chagas, CMV, are only excluded if they are being treated for active infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits Van Rhee, M.D., Phd, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ENK Cell Infusion
Started | 3
Completed | 1
Not Completed | 2
Not completed — Screen Failure | 2

BASELINE CHARACTERISTICS:
Population: Data includes only those participants that initiated study therapy.
Arm/Group | ENK Cell Infusion
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Increase in ENK (Expanded Natural Killer Cells) Cells 7 Days After Treatment
Description: Number of participants with at least 4 fold increase in absolute CD3-CD56+ NK cell count/uL blood 7 days after infusion over the pre-study baseline level
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | ENK Cell Infusion
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Arm/Group | ENK Cell Infusion
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENK Cell Infusion (N=1)
Grade 1 Anemia (Blood and lymphatic system disorders) | 1
Grade 2 Anemia (Blood and lymphatic system disorders) | 1
Grade 1 Arthritis (Musculoskeletal and connective tissue disorders) | 1
Grade 1 Bruising (Injury, poisoning and procedural complications) | 1
Grade 1 Cataract (Eye disorders) | 1
Grade 1 Constipation (Gastrointestinal disorders) | 1
Grade 1 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Grade 1 Edema-limb (General disorders) | 1
Grade 1 Hot Flashes (Vascular disorders) | 1
Grade 1 Hyperglycemia (Metabolism and nutrition disorders) | 1
Grade 1 Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Grade 1 Hyponatremia (Metabolism and nutrition disorders) | 1
Grade 3 Hyponatremia (Metabolism and nutrition disorders) | 1
Grade 1 Injection Site Reaction (General disorders) | 1
Grade 2 Injection Site Reaction (General disorders) | 1
Gade 1 Fatigue (General disorders) | 1
Grade 1 Pain - NOS (General disorders) | 1
Grade 1 Mood Alteration (Psychiatric disorders) | 1
Grade 1 Nausea (Gastrointestinal disorders) | 1
Grade 1 Neutropenia (Blood and lymphatic system disorders) | 1
Grade 2 Neutropenia (Blood and lymphatic system disorders) | 1
Grade 1 Pruritis (Skin and subcutaneous tissue disorders) | 1
Grade 1 Rigors/Chills (General disorders) | 1
Grade 1 SGOT (AST) Increase (Hepatobiliary disorders) | 1
Grade 1 SGPT (ALT) Increase (Hepatobiliary disorders) | 1
Grade 1 Thrombocytopenia (Blood and lymphatic system disorders) | 1
Grade 2 Thrombocytopenia (Blood and lymphatic system disorders) | 1
Grade 2 Leukopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes